CLINICAL TRIAL: NCT06578403
Title: Minimally Invasive Non-surgical Therapy Augmented With Internal Versus External Micro-needling in Treatment of Stage Iii Periodontitis: a Randomized Controlled Clinical Trial and Biochemical Trial
Brief Title: Effect of Internal and External Micro-needling in Treatment of Stage III Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Hasnaa Nassar abdelhamied ali, principle investigator, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MisrUST. MICRONEEDLE
Record Dates: First submitted 2024-07-07; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases
Keywords: microneedling; periodontitis; Minimally invasive non-surgical therapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: 1:1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator): minimally invasive non-surgical technique (MINST) in management of periodontitis stage III patients.
  Interventions: Other: minimally invasive non- surgical periodontal therapy
- external intervention (Experimental): minimally invasive non-surgical technique (MINST) with external microneedle (EMN) periodontitis stage III patients.
  Interventions: Device: external microneedling; Other: minimally invasive non- surgical periodontal therapy
- internal intervention (Experimental): minimally invasive non-surgical technique with an internal microneedle (IMN) on periodontitis stage III patients.
  Interventions: Other: minimally invasive non- surgical periodontal therapy; Device: internal micro_needling

INTERVENTIONS:
Device: external microneedling — external micro_needling
  Arms: external intervention
Other: minimally invasive non- surgical periodontal therapy — minimally invasive non- surgical periodontal therapy
Device: internal micro_needling — internal micro_ needling
  Arms: internal intervention

SUMMARY:
Periodontitis is a dysbiotic disease characterized by the destruction of the periodontium (alveolar bone, cementum, periodontal ligament, gingiva) and considered the main cause of tooth loss which is linked to a change in the microbial community from primarily beneficial bacteria, known as 'symbionts', to an imbalance with a high presence of harmful bacteria 'dysbiosis', also known as 'pathobionts'.

Ideally, periodontal therapy should eliminate inflammation, arrest the advancement of periodontal disease, enhance appearance, and create an environment conducive to health maintenance.Microneedling (MN) is known as "percutaneous collagen induction therapy." Micro injuries created by MN result in minimal superficial bleedings and create a wound-healing The body responds to micro-needling as if it's experiencing tissue trauma, leading to the release of various growth factors such as platelet-derived growth factors, transforming growth factors, connective tissue growth factors, and fibroblast growth factors. These growth factors induce the production of collagen to preserve skin integrity. After an injury, growth factors are released, promoting the proliferation of new cells. From day 5 to week 8, fibroblasts produce collagen and elastin fibers, thickening the tissue in a process known as neocollagenesis. Additionally, fibroblasts trigger neoangiogenesis by stimulating the proliferation of endothelial cells in the vessels. According to a randomized clinical trial comparing micro-needling and acellular dermal matrix, significant improvements were observed in various parameters(GT, RW, RD, CAL, PD, Rec- Red, and percentage of root coverage, with reduced PI and BOP at 3 and 6 months this study aim to The effect of minimally invasive non-surgical augmented with micro-needling, both externally and internally, for the management of stage III periodontitis

DETAILED DESCRIPTION:
Study Settings and Source of Patients The study will take place in the outpatient clinics of the oral medicine, periodontology, and Diagnosis department at the Faculty of Oral and Dental Surgery at Misr University for Science and Technology. All procedures will be conducted with the approval of the Research Ethics Committee (REC) of the Faculty of Oral and Dental Surgery at Misr University for Science and Technology.

SIX periodontitis stage III patients seeking periodontal therapy will be included in this study. The selection of patients will be done after careful clinical, radiographic, and periodontal examination according to the following inclusion and exclusion criteria.

Methods of measurement of outcome:

Clinical Parameters:

The following parameters will be recorded at baseline, 3 months after initial periodontal therapy and after 6 months.

1. Probing depth:

   UNC 15 probe will be used to measure the pocket depth from the gingival margin to the base of the pocket.
2. Gingival index [GI]:

   It is used to assess gingival inflammation .
3. Clinical attachment level [CAL]):

   Represents the extent of periodontal support that has been lost around a tooth and is measured with the periodontal probe as the distance from the cemento-enamel junction (CEJ) to the base of the pocket .
4. plaque index:

   The desirability of distinguishing clearly between the soft debris aggregates' severity and location.
5. Bleeding on probing POB:

   bleeding indices have been devised; some assess bleeding as simply present or absent, whereas others use grading in an attempt to assess severity of bleeding
6. Vas index :

A Visual Analogue Scale (VAS) is a pain rating scale 1,2,3,4,5,6,7,8,9 Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)

Biological assessment(Platelet-derived growth factor(PDGF) levels in gingival crevicular fluid Assessment of PDGF in gingival crevicular fluid at baseline,7,14 days

ELIGIBILITY:
Inclusion Criteria:

* Male or Female systematic health
* age ≥ 18 years
* Provide informed consent and willingness to cooperate with the study protocol.
* Periodontitis stage III patients:
* Probing depth≥6 mm
* CAL ≥5 mm.
* Radiographic bone loss (Extending to middle and beyond)
* Tooth loss ≥4 teeth.
* Each patient contributed a maximum of two sides.

Exclusion Criteria:

* smoker
* History of antibiotic in previous three months.
* Pregnant or lactating.
* Treatment with any systemic drug that influences the healing of hard and soft tissues.
* Patients who received periodontal treatment in the last 6 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Probing depth | 6month
  measure the pocket depth from the gingival margin to the base of the pocket using UNC 15 probe (mm)
Clinical attachment level [CAL]): | 6month
  measured with the periodontal probe as the distance from the cemento-enamel junction(CEJ) to the base of the pocket by UNC 15 probe (mm)
plaque index | 6 month
  The desirability of distinguishing clearly between the soft debris aggregates' severity and location by system Score 0 = The tooth surface is clean. - Score 1 = The tooth surface appears clean, but dental plaque can be removed from the gingival third with a sharp explorer. - Score 2 = Plaque is visible along the gingival margin. - Score 3 = The tooth surface is covered with abundant plaque
Bleeding on probing | 6 month
  bleeding indices have been devised; some assess bleeding as simply present or absent, whereas others use grading in an attempt to assess severity of bleeding is the score criteria: 0: no bleeding 1: one bleeding point appears 2: multiple bleeding points or one bleeding line appear 3: interdental triangle filled with blood 4: excessive bleeding when probing and blood flow to the marginal sulcus

SECONDARY OUTCOMES:
A Visual Analogue Scale (VAS) | immediately after phase 1 therapy
  a pain rating scale 1,2,3,4,5,6,7,8,9 Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)
Platelet-derived growth factor (PDGF) levels in gingival crevicular fluid | baseline,7,14 days.
  PDGF are major mitogens for many cell types of mesenchymal origin and for some cells that are neuroectodermal in origin, like oligodendrocytes. PDGF have chemoattractant properties and have been involved in bone formation, erythropoiesis, wound healing and angiogenesis
crestal bone level | after 6 month
  assessment of crestal bone level by periapical x-ray